CLINICAL TRIAL: NCT03087890
Title: Randomized Clinical Trial to Assess Whether the Duration of Cotrimoxazole Preventive Therapy in HIV Patients With CD4 Counts >350 CD4 Cells/µL by Antiretroviral Treatment Influences the Rate of Carriage of Multidrug-resistant Bacteria
Brief Title: Impact of Cotrimoxazole Use in Immunocompetent HIV Patients on Carriage of Antimicrobial Resistant Bacteria
Acronym: CoTrimResist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Muhimbili University of Health and Allied Sciences (Other); Helse Vest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REK2015/540; TZ16CT007 (Other: Tanzania Food and Drugs Authority); NIMRlHQ/R.SaJVol. 1X12144 (Other: National Institute for Medical Research, Tanzania); 2015-10-27/AEC/Vol.X/54 (Other: Muhimbili University of Health and Allied Sciences); REK2015/540 (Other: Regional Committee for Medical Ethics, Western Norway)
Record Dates: First submitted 2017-03-08; First posted 2017-03-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: HIV-1-infection; Pneumocystis Pneumonia; Opportunistic Infections; Preventive Therapy; Antibiotic Side Effect
Keywords: Microbial drug resistance; Beta-lactamase; Cotrimoxazole; Trimethoprim-sulfamethoxazole; Tanzania
MeSH Terms: conditions — Pneumonia, Pneumocystis; Opportunistic Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed hiv-1 infection and good immunological status defined as CD4 counts of >350 pr microliter, will be randomised to receive cotrimoxazole (160mg/800mg) daily or placebo for 48 weeks. Rectal and nasal swabs will be collected on day 0, 14, week 24 and week 48. The swabs will be analysed for the presence of bacterial species with focus on certain multidrug-resistant bacteria such as ESBL (extended spectrum beta-lactamase)-producing Gram negative bacteria, MRSA (methicillin-resistant Staphylococcus aureus) and VRE (Vancomycin-resistant enterococci). Patients will also be monitored closely on monthly visits to assess for any adverse events.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients in one study arm will receive 2 tablets daily of Cotrimoxazole (trimethoprim 80mg + sulfamethoxazole 400mg), these tablets are purchased locally in Tanzania, and are the same as used for pneumocystis preventive therapy under the National AIDS control programme. Participants in arm 2 will receive 2 placebo tablets daily. These tablets have been manufactured by Kragero Tablettproduksjon AS, Norway, and care has been taken to make them look as similar as possible to the locally purchased cotrimoxazole tablets from Tanzania. Neither study participants, care providers, investigators or outcome assessors will know which patients receive cotrimoxazole or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cotrimoxazole (Active Comparator): Patients in the Cotrimoxazole study arm will receive 2 tablets daily of Cotrimoxazole (trimethoprim 80mg + sulfamethoxazole 400mg), these tablets are purchased locally in Tanzania, and are the same as used for pneumocystis preventive therapy under the National AIDS control programme.
  Interventions: Drug: Cotrimoxazole
- Placebo (Placebo Comparator): Participants in the Placebo arm will receive 2 placebo tablets daily. These tablets have been manufactured by Kragero Tablettproduksjon AS, Norway, and care has been taken to make them look as similar as possible to the locally purchased cotrimoxazole tablets from Tanzania. Neither study participants, care providers, investigators or outcome assessors will know which patients receive cotrimoxazole or placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cotrimoxazole — Patients will receive preventive treatment with 2 tablets cotrimoxazole (80 mg trimethoprim, 400mg sulfamethoxazole) daily for 48 weeks
  Other Names: Trimethoprim - sulfamethoxazole
  Arms: Cotrimoxazole
Drug: Placebo — Patients will receive 2 tablets placebo daily for 48 weeks
  Other Names: Placebo tablet with no active drug
  Arms: Placebo

SUMMARY:
Cotrimoxazole preventive therapy (CPT) is recommended for prevention of morbidity and mortality due to Pneumocystis pneumonia and other infections in HIV positive patients with low immunity. Common clinical practice is to start CPT in any patient with CD4 counts below 200/µL, and, conversely, to stop CPT when immunity has been restored by antiretroviral treatment to CD4 counts above 200/µL or when viral suppression has been documented for 3 months. However, the latest WHO guidelines widely expands the indication for CPT by advocating for settings with high prevalence of malaria and bacterial infections, that all patients with HIV start CPT regardless of CD4 counts and clinical stage. Furthermore, WHO recommends these patients to continue CPT indefinitely regardless of evidence of immune restoration (The recommendation is for settings with high prevalence of malaria and bacterial infections, not for high-income countries). There is limited scientific evidence to recommend prolonged CPT, as studies have shown it is associated with modestly reduced morbidity due to pneumonia, meningitis and malaria, but no corresponding reduction in mortality. The impact of such a large increase in antibiotic use on the emergence of antimicrobial resistance has not been thoroughly considered. Our previous studies in Tanzania showed that multidrug-resistant bacteria frequently cause bloodstream infections with resultant very high case-fatality rates. As genes encoding for multiple antibiotic resistance traits are transferred by plasmids together with resistance towards cotrimoxazole, prolonged CPT will likely favor the selection of carriage of multidrug-resistant gut bacteria. The proposed randomized clinical trial is designed to assess whether prolonged CPT in HIV-positive patients results in increased fecal carriage of multi-drug resistant gut microbes or increased nasal carriage of methicillin-resistant Staphylococcus aureus (MRSA). Secondary endpoints are morbidity (clinical events, hospitalizations) and mortality. Stool specimens, nasal swabs and clinical data will be collected from persons attending voluntary counseling and testing facilities and HIV-clinics in Dar es Salaam, Tanzania. The study results may have important impact on public health in terms of assisting development of rational recommendations for CPT use, and may help prevent emerging antibiotic resistance.

DETAILED DESCRIPTION:
Background Bacterial infections account for a large proportion of global morbidity and mortality. While antimicrobial drugs have helped save millions from the consequences of these infections, emerging antimicrobial resistance now threatens to reverse those gains. The HIV-epidemic renders large populations drastically more susceptible to bacterial infections, particularly in Sub-Saharan Africa, where HIV is rampant and health-systems to deal with the consequences are insufficient. Indiscriminate use of antimicrobials is thought to be the main driving force behind emerging resistance. The opportunistic infection Pneumocystis jirovecii pneumonia (PJP) is a major cause of mortality among HIV-infected people with low immunity. Continuous cotrimoxazole preventive therapy (CPT) has proved to reduce morbidity and mortality from PJP globally, as well as in Africa where the burden of HIV is largest. The impact of this large-scale antibiotic use on emergence of antimicrobial resistance in Africa remains unclear. In a recent literature review, Sibanda and colleagues found only two studies specifically designed to answer the question of whether CPT induced resistance in common bacterial pathogens, and 15 other studies that assessed the question as sub-analyses of studies designed for other purposes. The two targeted studies both assessed resistance in pneumococci, one finding increased resistance to clindamycin in the CPT group, neither finding any difference in resistance to penicillin. While most of the other 15 studies assessed penicillin-resistance in pneumococci and methicillin-resistance in Staphylococcus aureus (MRSA), only two studies evaluated the effect on Gram-negative bacteria. Among these, the study from San Francisco showed significantly higher temporal increase from 1988 to 1995 in resistance to cotrimoxazole, ampicillin, cefazolin and gentamicin in clinical isolates of E. coli from HIV-positives than from HIV-negatives. The study of HIV-infected children with pneumonia in Cape Town did not find any association between CPT and resistance in clinical isolates, including 26 isolates of Klebsiella pneumonia, the most prevalent Gram-negative microbe in this study. In previous research in Tanzania, we found that multi-drug resistance in Gram-negative bacteria is prevalent and a problem of major public health concern, as invasive infections with such bacteria was associated with a large increase in mortality. Our study found case-fatality rates (>70%) approaching those of the pre-antibiotic era in systemic bacterial infections with multi-resistant Gram-negative bacteria harboring extended-spectrum beta-lactamase (ESBL) resistance. ESBLs are enzymes that render the all-important antibiotics, penicillins and cephalosporins, useless. We also confirmed previous findings that case-fatality rates from bacterial sepsis was higher in HIV-infected than HIV-negative patients. Most disturbingly, our study confirmed that in multidrug-resistant Gram-negative bacteria the gene encoding for ESBL resistance was transferred by plasmids together with resistance to several other antibiotics, including cotrimoxazole. Thus, it is plausible that widespread cotrimoxazole use could lead to selection of multidrug-resistant Gram-negative bacteria in the gut of HIV-patients, which consequently could contribute to the rapid spread of these harmful and difficult-to-treat bacteria. In high-resource countries, it has been shown that CPT can safely be discontinued when CD4 counts increase beyond 200/uL. Recent studies from Sub-Saharan Africa indicate that prolonged CPT after immune restoration to CD4 counts > 200/µL by antiretroviral treatment (ART) may be beneficial as it is associated with reduced hospitalization from malaria and bacterial infections in children. There was, however, no difference in mortality among those who stopped and continued CPT. In the "2014 supplement to the WHO guidelines on the use of antiretroviral drugs for treating and preventing HIV infection", the recommendation for CPT use is widely expanded for settings with high prevalence of malaria and bacterial infections, where it is recommended that all patients with HIV start CPT regardless of CD4 counts and clinical stage and receive prolonged CPT for indefinitely time. Tanzanian national guidelines recommend discontinuing CPT when patients are stabilized with CD4 counts >350/µL, which is a more extensive recommendation than European guidelines, but much less extensive than the WHO recommendations for "settings with high prevalence of malaria and bacterial infections".

Cotrimoxazole has been widely used for a number of different indications and, as a result, cotrimoxazole resistance in general has increased. Given the limited published data on these important public health issues, we designed this study to address the potential impact of prolonged CPT on antimicrobial resistance development with particular focus on Gram-negative gut microbes, VRE (vancomycin-resistant enterococci), and nasal carriage of MRSA. If the study should confirm a marked increase in carriage of multidrug-resistant bacteria in patients on prolonged CPT this needs to be considered when developing new guidelines. We also aim at assessing whether restoration of immunity by ART could be a way to counteract this threat of antimicrobial resistance. This proposed randomized clinical trial will be performed in the setting of the ongoing Dar es Salaam - Bergen collaborative initiative and will include local investigators and laboratory workers, along with Norwegian investigators with scientific experience from clinical and molecular studies in Tanzania.

Problem statement/ research gap CPT has been standard of care for preventing PJP and other infections among HIV-infected patients with CD4 counts < 200µL since the early 1990s. The recent recommendation by WHO to give CPT indefinitely to HIV-infected people in resource-constrained settings, even to those with initial good immunity (CD4 counts above 350/µL) and to those whose immunity has been restored by antiretroviral treatment, would lead to a massive increase in cotrimoxazole consumption in Sub-Saharan Africa, which has the largest burden of HIV-infection. While this recommendation is based on limited scientific data regarding short-term morbidity, there is no evidence of improved survival and the potential harmful implication for selection of multidrug-resistant bacteria in HIV-patients on prolonged CPT has not been comprehensively studied.

Rationale of the study Continuing CPT indefinitely stable good immunity with CD4 counts >350/µL has been shown to reduce morbidity, but not mortality, in persons living with HIV in resource-constrained settings. Complying with recommendation for continuation of CPT indefinitely in patients with restored immunity and virological control would imply a massively increased consumption of cotrimoxazole in HIV-endemic countries. The risk of increased carriage of multidrug-resistant bacteria among HIV-patients on prolonged CPT has not been comprehensively studied, but has potentially grave implications for public health, since systemic infections with these resistant bacteria are very difficult to treat and associated with very high mortality rates. The current study is designed to assess whether prolonged CPT is associated with increased carriage of multidrug-resistant bacteria. The results of this study may have important implications for development of new guidelines on CPT use for resource-constrained settings and may help preventing emerging antibacterial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who provide written informed consent will be included
* Patients aged 18 years or older with newly diagnosed HIV-infection and CD4 counts of ≥ 350 per microliter will be included for randomisation to receive placebo or cotrimoxazole preventive treatment.
* Persons testing hiv negative at the participating clinics will be included as additional control group but not randomised to interventions
* Persons testing hiv-positive and having impaired immunity with CD4 count below will be included as additional control group but not randomised for intervention. This group will routinely receive cotrimoxazole prophylaxis from the national AIDS control program, and not followed-up further in this study.

Exclusion Criteria:

* CD4<350 per microliter at enrollment
* Patients allergic to cotrimoxazole
* Children under age of 18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Change in carriage of resistant bacteria in gut and/or nose by week 2 | From baseline to day 14
  Change in the proportion who carry antibiotic-resistant bacteria, including presence of extended-spectrum beta-lactamase (ESBL) producing gram-negative bacteria or vancomycin-resistant enterococci (VRE) on microbiological examination of fecal swab, or methicillin-resistant Staphylococcus aureus (MRSA) on microbiological examination of nasal swab, from baseline to day 14
Change in carriage of resistant bacteria in gut and/or nose by week 24 | From baseline to week 24
  Change in the proportion who carry antibiotic-resistant bacteria, including presence of extended-spectrum beta-lactamase (ESBL) producing gram-negative bacteria or vancomycin-resistant enterococci (VRE) on microbiological examination of fecal swab, or methicillin-resistant Staphylococcus aureus (MRSA) on microbiological examination of nasal swab, from baseline to week 24
Change in carriage of resistant bacteria in gut and/or nose by week 48 | From baseline to week 48
  Change in the proportion who carry antibiotic-resistant bacteria, including presence of extended-spectrum beta-lactamase (ESBL) producing gram-negative bacteria or vancomycin-resistant enterococci (VRE) on microbiological examination of fecal swab, or methicillin-resistant Staphylococcus aureus (MRSA) on microbiological examination of nasal swab, from baseline to week 48

SECONDARY OUTCOMES:
Adverse events | From baseline to 48 weeks
  Adverse events graded as a) light, b) moderate, c) severe, d) life-threatening or e) fatal will be registered through patients' monthly visits to clinic and additional follow-up as required
Mortality | From baseline to 48 weeks
  All cause mortality
Morbidity | From baseline to 48 weeks
  Documented episode of malaria, pneumonia, diarrhea and hospital admission

OTHER OUTCOMES:
Difference in carriage of resistant bacteria in gut and/or nose between HIV positive patients and HIV negative controls | At baseline
  Difference in the proportion who carry antibiotic-resistant bacteria, including presence of extended-spectrum beta-lactamase (ESBL) producing gram-negative bacteria or vancomycin-resistant enterococci (VRE) on microbiological examination of fecal swab, or methicillin-resistant Staphylococcus aureus (MRSA) on microbiological examination of nasal swab, between HIV positive patients and HIV negative controls
Difference in carriage of resistant bacteria in gut and/or nose between HIV positive patients with CD4 counts above and below 350 | At baseline
  Difference in the proportion who carry antibiotic-resistant bacteria, including presence of extended-spectrum beta-lactamase (ESBL) producing gram-negative bacteria or vancomycin-resistant enterococci (VRE) on microbiological examination of fecal swab, or methicillin-resistant Staphylococcus aureus (MRSA) on microbiological examination of nasal swab, between HIV positive patients with CD4 counts above and below 350

CONTACTS AND LOCATIONS:
Overall Officials: Joel Manyahi, MD, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (6):
- Tanzania (6):
  - Amana Regional Referral Hospital, Dar es Salaam
  - Mbagala District Hospital, Dar es Salaam
  - Mnazimmoja Health Centre, Dar es Salaam
  - Mwananyamala Regional Referral Hospital, Dar es Salaam
  - Pasada Upendano, Dar es Salaam
  - Temeke Regional Referral Hospital, Dar es Salaam

IPD SHARING:
Plan to Share IPD: Undecided
There are currently no plans for sharing data with other researchers.

REFERENCES:
- [Background] Anglaret X, Chene G, Attia A, Toure S, Lafont S, Combe P, Manlan K, N'Dri-Yoman T, Salamon R. Early chemoprophylaxis with trimethoprim-sulphamethoxazole for HIV-1-infected adults in Abidjan, Cote d'Ivoire: a randomised trial. Cotrimo-CI Study Group. Lancet. 1999 May 1;353(9163):1463-8. doi: 10.1016/s0140-6736(98)07399-1. PMID 10232311
- [Background] Mermin J, Lule J, Ekwaru JP, Malamba S, Downing R, Ransom R, Kaharuza F, Culver D, Kizito F, Bunnell R, Kigozi A, Nakanjako D, Wafula W, Quick R. Effect of co-trimoxazole prophylaxis on morbidity, mortality, CD4-cell count, and viral load in HIV infection in rural Uganda. Lancet. 2004 Oct 16-22;364(9443):1428-34. doi: 10.1016/S0140-6736(04)17225-5. PMID 15488218
- [Background] Sibanda EL, Weller IV, Hakim JG, Cowan FM. Does trimethoprim-sulfamethoxazole prophylaxis for HIV induce bacterial resistance to other antibiotic classes? Results of a systematic review. Clin Infect Dis. 2011 May;52(9):1184-94. doi: 10.1093/cid/cir067. PMID 21467024
- [Background] Hamel MJ, Greene C, Chiller T, Ouma P, Polyak C, Otieno K, Williamson J, Shi YP, Feikin DR, Marston B, Brooks JT, Poe A, Zhou Z, Ochieng B, Mintz E, Slutsker L. Does cotrimoxazole prophylaxis for the prevention of HIV-associated opportunistic infections select for resistant pathogens in Kenyan adults? Am J Trop Med Hyg. 2008 Sep;79(3):320-30. PMID 18784222
- [Background] Gill CJ, Mwanakasale V, Fox MP, Chilengi R, Tembo M, Nsofwa M, Chalwe V, Mwananyanda L, Mukwamataba D, Malilwe B, Champo D, Macleod WB, Thea DM, Hamer DH. Effect of presumptive co-trimoxazole prophylaxis on pneumococcal colonization rates, seroepidemiology and antibiotic resistance in Zambian infants: a longitudinal cohort study. Bull World Health Organ. 2008 Dec;86(12):929-38. doi: 10.2471/blt.07.049668. PMID 19142293
- [Background] Martin JN, Rose DA, Hadley WK, Perdreau-Remington F, Lam PK, Gerberding JL. Emergence of trimethoprim-sulfamethoxazole resistance in the AIDS era. J Infect Dis. 1999 Dec;180(6):1809-18. doi: 10.1086/315132. PMID 10558935
- [Background] Zar HJ, Hanslo D, Hussey G. The impact of HIV infection and trimethoprim-sulphamethoxazole prophylaxis on bacterial isolates from children with community-acquired pneumonia in South Africa. J Trop Pediatr. 2003 Apr;49(2):78-83. doi: 10.1093/tropej/49.2.78. PMID 12729288
- [Background] Blomberg B, Mwakagile DS, Urassa WK, Maselle SY, Mashurano M, Digranes A, Harthug S, Langeland N. Surveillance of antimicrobial resistance at a tertiary hospital in Tanzania. BMC Public Health. 2004 Oct 11;4:45. doi: 10.1186/1471-2458-4-45. PMID 15476559
- [Background] Blomberg B, Jureen R, Manji KP, Tamim BS, Mwakagile DS, Urassa WK, Fataki M, Msangi V, Tellevik MG, Maselle SY, Langeland N. High rate of fatal cases of pediatric septicemia caused by gram-negative bacteria with extended-spectrum beta-lactamases in Dar es Salaam, Tanzania. J Clin Microbiol. 2005 Feb;43(2):745-9. doi: 10.1128/JCM.43.2.745-749.2005. PMID 15695674
- [Background] Blomberg B, Manji KP, Urassa WK, Tamim BS, Mwakagile DS, Jureen R, Msangi V, Tellevik MG, Holberg-Petersen M, Harthug S, Maselle SY, Langeland N. Antimicrobial resistance predicts death in Tanzanian children with bloodstream infections: a prospective cohort study. BMC Infect Dis. 2007 May 22;7:43. doi: 10.1186/1471-2334-7-43. PMID 17519011
- [Background] Tellevik MG, Sollid JE, Blomberg B, Jureen R, Urassa WK, Langeland N. Extended-spectrum beta-lactamase-type SHV-12-producing Enterobacteriaceae causing septicemia in Tanzanian children: vectors for horizontal transfer of antimicrobial resistance. Diagn Microbiol Infect Dis. 2007 Nov;59(3):351-4. doi: 10.1016/j.diagmicrobio.2007.06.015. Epub 2007 Sep 18. PMID 17878065
- [Background] Furrer H, Opravil M, Rossi M, Bernasconi E, Telenti A, Bucher H, Schiffer V, Boggian K, Rickenbach M, Flepp M, Egger M; Swiss HIV Cohort Study. Discontinuation of primary prophylaxis in HIV-infected patients at high risk of Pneumocystis carinii pneumonia: prospective multicentre study. AIDS. 2001 Mar 9;15(4):501-7. doi: 10.1097/00002030-200103090-00009. PMID 11242147
- [Background] Bwakura-Dangarembizi M, Kendall L, Bakeera-Kitaka S, Nahirya-Ntege P, Keishanyu R, Nathoo K, Spyer MJ, Kekitiinwa A, Lutaakome J, Mhute T, Kasirye P, Munderi P, Musiime V, Gibb DM, Walker AS, Prendergast AJ. A randomized trial of prolonged co-trimoxazole in HIV-infected children in Africa. N Engl J Med. 2014 Jan 2;370(1):41-53. doi: 10.1056/NEJMoa1214901. PMID 24382064
- [Background] Zachariah R, Harries AD, Spielmann MP, Arendt V, Nchingula D, Mwenda R, Courtielle O, Kirpach P, Mwale B, Salaniponi FM. Changes in Escherichia coli resistance to co-trimoxazole in tuberculosis patients and in relation to co-trimoxazole prophylaxis in Thyolo, Malawi. Trans R Soc Trop Med Hyg. 2002 Mar-Apr;96(2):202-4. doi: 10.1016/s0035-9203(02)90306-8. PMID 12055816
- [Derived] Manyahi J, Moyo SJ, Langeland N, Blomberg B. Genetic determinants of macrolide and tetracycline resistance in penicillin non-susceptible Streptococcus pneumoniae isolates from people living with HIV in Dar es Salaam, Tanzania. Ann Clin Microbiol Antimicrob. 2023 Feb 20;22(1):16. doi: 10.1186/s12941-023-00565-3. PMID 36803640
- [Derived] Manyahi J, Moyo SJ, Aboud S, Langeland N, Blomberg B. Predominance of PVL-negative community-associated methicillin-resistant Staphylococcus aureus sequence type 8 in newly diagnosed HIV-infected adults, Tanzania. Eur J Clin Microbiol Infect Dis. 2021 Jul;40(7):1477-1485. doi: 10.1007/s10096-021-04160-2. Epub 2021 Feb 14. PMID 33586013
- [Derived] Manyahi J, Moyo S, Aboud S, Langeland N, Blomberg B. High rate of antimicrobial resistance and multiple mutations in the dihydrofolate reductase gene among Streptococcus pneumoniae isolated from HIV-infected adults in a community setting in Tanzania. J Glob Antimicrob Resist. 2020 Sep;22:749-753. doi: 10.1016/j.jgar.2020.06.026. Epub 2020 Jul 9. PMID 32653726